CLINICAL TRIAL: NCT00524160
Title: Open-Label Study To Assess The Effect On Pain Control Of Durogesic (Fentanyl Transdermic Therapeutic System) Treatment In Subjects With Rheumatoid Arthritis Or Osteoarthritis Of The Knee Or Hip.
Brief Title: A Study of the Effect on Pain Control of Treatment With Fentanyl, Administered Through the Skin, in Patients With Rheumatoid Arthritis or Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR001981
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Arthritis; Osteoarthritis; Rheumatoid Arthritis
Keywords: Fentanyl; opioid analgesics; arthritis; osteoarthritis; rheumatoid arthritis; transdermal administration
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid

INTERVENTIONS:
Drug: Fentanyl transdermal patch

SUMMARY:
The purpose of this study is to assess the degree of pain control achieved by treatment with fentanyl, administered via adhesive patches applied to the skin ('transdermal system") in patients with rheumatoid arthritis or osteoarthritis of the knee or hip. Treatment will be administered fo r4 weeks, added on to existing therapy with other medications.

DETAILED DESCRIPTION:
Chronic, non-cancer pain may result from injury or illness, such as rheumatoid arthritis or osteoarthritis, which causes suffering and a reduction in the quality of life. Opioids, such as fentanyl, are beneficial as potent pain-relieving drugs in patients with continuous pain. This is an open-label, prospective study to assess the degree of pain control provided by treatment with fentanyl administered through the skin via adhesive patches ("transdermal system") for 28 days in patients with rheumatoid arthritis or osteoarthritis of the hip or knee, whose pain is inadequately controlled by other medications. During the first week of treatment, a prophylactic anti-nausea and vomiting agent will be given to patients to control these symptoms that can occur during opioid therapy. After 28 days, patients who do not respond adequately to treatment will be tapered off by gradually reducing the dose of fentanyl. Assessment of effectiveness will include a rating of pain control (excellent, good, moderate, poor, very poor), Pain Assessment Questionnaire, Quality of Life Questionnaire (SF-36), Health Assessment Questionnaire (HAQ), recording of the usage of any additional pain-relieving medications, and an evaluation of the anti-nausea and vomiting treatment. Safety evaluations include incidence of adverse events, and physical examinations. The study hypothesis is that patients with rheumatoid arthritis or osteoarthritis of the hip or knee whose pain is not adequately controlled by other medications will show an improvement in pain control after 28 days of treatment with the fentanyl transdermal system. Fentanyl transdermal patches to deliver from 25 micrograms/hr to 100 micrograms/hr, changed every 3 days, for 28 days; doses may be adjusted for adequate pain control, Anti-nausea tablets (Metoclopramide, 10 mg, 3 times/day) during first week. Paracetamol tablets (500mg) to supplement pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the American College of Rheumatology criteria for rheumatoid arthritis (RA) or osteoarthritis (OA) of the hip or knee and have moderate or severe pain that is not adequately controlled by other medications (paracetamol (acetaminophen), NSAIDs, COX-2 inhibitors, weak opioids)
* OA patients must be in need of and waiting for hip or knee replacement
* RA patients using disease modifying antirheumatic drugs (DMARDs) must have been on stable dose of medication for >=3 months.

Exclusion Criteria:

* Patients who have received regular treatment with strong opioids during the month prior to study
* another continuous pain that stands out compared to RA or OA pain
* skin disease or known allergy or hypersensitivity to fentanyl or to the adhesives
* history of liver disease
* new physical therapy or change in that therapy within one month of study
* pregnant or nursing females, or those without adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2001-07; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Assessment of pain control (excellent, good, moderate, poor, very poor) and Pain Assessment Questionnaire at baseline and then weekly through Day 28.

SECONDARY OUTCOMES:
Incidence of adverse events throughout study; efficacy of anti-nausea treatment (weekly); SF-36 Quality of Life Questionnaire and Health Assessment Questionnaire (HAQ) at start of treatment and Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Pavelka K, Le Loet X, Bjorneboe O, Herrero-Beaumont G, Richarz U. Benefits of transdermal fentanyl in patients with rheumatoid arthritis or with osteoarthritis of the knee or hip: an open-label study to assess pain control. Curr Med Res Opin. 2004 Dec;20(12):1967-77. doi: 10.1185/030079904X14120. PMID 15701214
- [Result] Herrero-Beaumont G, Bjorneboe O, Richarz U. Transdermal fentanyl for the treatment of pain caused by rheumatoid arthritis. Rheumatol Int. 2004 Nov;24(6):325-32. doi: 10.1007/s00296-004-0520-7. Epub 2004 Oct 5. PMID 15480678
- [Result] Le Loet X, Pavelka K, Richarz U. Transdermal fentanyl for the treatment of pain caused by osteoarthritis of the knee or hip: an open, multicentre study. BMC Musculoskelet Disord. 2005 Jun 15;6:31. doi: 10.1186/1471-2474-6-31. PMID 15958159